CLINICAL TRIAL: NCT01797276
Title: Dichloroacetate Treatment of Congenital Lactic Acidosis Phase B: Expanded Access
Acronym: CLA
Status: No longer available | Type: Expanded Access
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB#420-2005
Record Dates: First submitted 2013-02-15; First posted 2013-02-22 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Mitochondrial Enzyme Deficiencies
Keywords: Dichloroacetate (DCA); Congenital Lactic Acidosis (CLA); acidosis; orphan disease
MeSH Terms: conditions — Acidosis; Rare Diseases | interventions — Dichloroacetic Acid

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: Dichloroacetate — Subjects are given DCA 25mg/kg in a divided dose twice a day.
  Other Names: DCA

SUMMARY:
Expanded access to DCA as continued treatment for congenital lactic acidosis.

DETAILED DESCRIPTION:
Subjects who participated in a Phase 3 Randomized Controlled Trial of DCA for treatment of Congenital Lactic Acidosis (CLA) are eligible to continue treatment with investigational medication DCA at the same dose of 25mg/kg/day for expanded access. Study participants must travel to the study site for bi-annual evaluation by the study investigator. Bi-annual evaluation will include an interim medical history review, physical exam, blood collection for DCA trough level, and urine pregnancy testing (if indicated).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital lactic acidosis
* Participation in Study: #183-1992: Dichloroacetate Treatment of Congenital Lactic Acidosis Exclusion Criteria:
* Intolerance to DCA

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Peter W. Stacpoole, PhD, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Box 100226, Gainesville, Florida, United States